CLINICAL TRIAL: NCT02265965
Title: Randomized Controlled Trial of IV Nitroglycerin in Cesarean Deliveries After Second Stage Arrest for the Prevention of Uterine Extension
Brief Title: Trial of IV NTG for CD After Second Stage Arrest for the Prevention of Uterine Extension
Acronym: NITRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCSF-OB-NTG
Record Dates: First submitted 2014-09-22; First posted 2014-10-16 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Prolonged Second Stage of Labor

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous Nitroglycerin (Experimental): Subjects will receive IV nitroglycerin at the time of Hysterotomy. Infusion will be stopped once neonate is delivered
  Interventions: Drug: intravenous nitroglycerin
- Intravenous Saline (No Intervention): Subjects will receive IV saline at the time of Hysterotomy. Infusion will be stopped once neonate is delivered

INTERVENTIONS:
Drug: intravenous nitroglycerin — Infusion at started at time of hysterotomy and stopped at neonate delivery
  Arms: Intravenous Nitroglycerin

SUMMARY:
Randomized controlled clinical trial of IV nitroglycerin at cesarean delivery for second stage arrest of descent to prevent or uterine extension at the hysterectomy site.

DETAILED DESCRIPTION:
Intravenous nitroglycerin resulting in uterine relaxation has been standardly utilized for various obstetrics conditions, e.g. breech extraction of second twin in vaginal deliveries, uterine relaxation after tachysystole in labor, prior to external cephalic version, and during difficult fetal extraction during cesarean delivery for arrest of descent in labor. Currently the use of nitroglycerin is at equipoise in obstetrics for difficult cesarean delivery after second stage arrest in labor. The clinical trial will randomize women who undergo cesarean delivery for second stage arrest in labor to receive IV nitroglycerin vs saline at the time of hysterotomy. The primary outcomes will be maternal: uterine extension, blood loss, total fetal extraction time, surgical time; neonatal: cord gases at delivery, apgar scores, admission to neonatal intensive care unit.

ELIGIBILITY:
Inclusion Criteria: women 37weeks or greater gestation diagnosed with second stage arrest of descent undergoing cesarean delivery -

Exclusion Criteria: elective, active phase arrest cesarean delivery, successful operative vaginal delivery

-

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Lucero, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University California San Francisco-Labor and Delivery, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Isquick S, Henry D, Nakagawa S, Moghadassi M, Thiet MP, Norton M, Lucero J. The association between nitroglycerin use and adverse outcomes in women undergoing cesarean delivery in the second stage of labor. J Matern Fetal Neonatal Med. 2017 Jun;30(11):1297-1301. doi: 10.1080/14767058.2016.1212010. Epub 2016 Aug 2. PMID 27405400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Nitroglycerin | Intravenous Saline
Started | 7 | 11
Completed | 7 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Nitroglycerin | Intravenous Saline | Total
Number analyzed (Participants) | 7 | 11 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 11 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (4.1) | 34.3 (3.3) | 34.7 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 11 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 8 | 11
  Black | 0 | 1 | 1
  Asian/Pacific Islander | 3 | 2 | 5
  Hispanic | 0 | 0 | 0
  Multi-racial or other | 1 | 0 | 1
Maternal body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.4 (3.9) | 25.3 (4.2) | 24.2 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Uterine Extension of Hysterotomy
Description: Obstetrician determined whether the subject had an uterine extension.
Time Frame: During cesarean delivery, estimated to be within 4 hours after diagnosis of second stage arrest
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Nitroglycerin | Intravenous Saline
Number analyzed (Participants) | 7 | 11
Participants | 3 | 4

2. Primary Outcome: Umbilical Artery Blood pH
Description: Measure of umbilical artery blood pH
Time Frame: At time of cesarean delivery, estimated to be within 4 hours after diagnosis of second stage arrest
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Intravenous Nitroglycerin | Intravenous Saline
Number analyzed (Participants) | 7 | 11
pH | 7.3 (0) | 7.3 (0)

3. Primary Outcome: Number of Participants With Deliveries After Which Neonate is Admitted to NICU
Time Frame: After cesarean delivery, estimated to be within 4 hours after diagnosis of second stage arrest
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Nitroglycerin | Intravenous Saline
Number analyzed (Participants) | 7 | 11
Participants | 1 | 2

4. Primary Outcome: Number of Participants With Deliveries in Which Cord Blood Base Deficit is More Negative Than or Equal to Negative 12
Description: A cord blood base deficit more negative than negative 12 is abnormal and a sign of metabolic acidosis.
Time Frame: At time of cesarean delivery, estimated to be within 4 hours after diagnosis of second stage arrest
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Nitroglycerin | Intravenous Saline
Number analyzed (Participants) | 7 | 11
Participants | 7 | 11

5. Primary Outcome: APGAR at 5 Minutes
Description: The APGAR scale is determined by evaluating the newborn baby on five simple criteria -- Appearance, Pulse, Grimace, Activity, Respiration -- on a scale from zero to two, then summing up the five values thus obtained. The resulting APGAR score ranges from zero to 10. Zero is the worst possible score and 10 is the highest possible score.
Time Frame: Immediately after cesarean delivery, estimated to be within 4 hours after diagnosis of second stage arrest
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Nitroglycerin | Intravenous Saline
Number analyzed (Participants) | 7 | 11
score on a scale | 9 [9 to 9] | 9 [8 to 9]

6. Secondary Outcome: Fetal Extraction Time in Seconds
Description: Time from uterine incision to delivery (body of neonate fully extracted from uterus)
Time Frame: At time of cesarean delivery, estimated to be within 4 hours after diagnosis of second stage arrest
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intravenous Nitroglycerin | Intravenous Saline
Number analyzed (Participants) | 7 | 11
seconds | 104.9 (33.1) | 131 (84.1)

7. Secondary Outcome: Total Operative Time in Minutes
Description: Time from uterine incision to out of room
Time Frame: After cesarean delivery, estimated to be within 4 hours after diagnosis of second stage arrest
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intravenous Nitroglycerin | Intravenous Saline
Number analyzed (Participants) | 7 | 11
minutes | 68.3 (22.0) | 74.2 (21.1)

8. Secondary Outcome: Surgical Blood Loss
Description: Total blood loss will be measured
Time Frame: During and after cesarean delivery, estimated to be within 4 hours after diagnosis of second stage arrest
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Intravenous Nitroglycerin | Intravenous Saline
Number analyzed (Participants) | 7 | 11
ml | 935.7 (217.4) | 1036.4 (201.4)

ADVERSE EVENTS:
Time Frame: Adverse event data were evaluated at 6 months.
Arm/Group | Intravenous Nitroglycerin | Intravenous Saline
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/11
Other Adverse Events (participants affected / at risk) | 0/7 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT02265965/Prot_SAP_000.pdf